CLINICAL TRIAL: NCT02800915
Title: Telemedicine Makes the Patient Stay in Hospital at Home. Service Innovation With Focus on Multidisciplinary Collaboration
Brief Title: Telemedicine Makes the Patient Stay in Hospital at Home
Acronym: TeleSCIpi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnaas Rehabilitation Hospital (Other)
Collaborators: Haukeland University Hospital (Other); University of Oslo (Other); Central Jutland Regional Hospital (Other); Sahlgrenska University Hospital (Other); Oslo University Hospital (Other); University Hospital of Trondheim, Norway (Unknown); Oslo Centre for Biostatistics and Epidemiology, Norway (Unknown); Norwegian Centre for Integrated Care and Telemedicine (NST), Norway (Unknown); Rigshospitalet, Denmark (Other); University of Alabama at Birmingham (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ingebjørg Irgens, MD-PRM/ PhD- candidate, Sunnaas Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/684
Record Dates: First submitted 2016-05-05; First posted 2016-06-15 (Estimated); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Spinal Cord Injury; Pressure Injury
Keywords: Spinal Cord Injury; Pressure Injury; Health Related Quality of Life; Telemedicine; Service Innovation; Rehabilitation; Interdisciplinary collaboration; User-participation; Activity and participation; Health economics
MeSH Terms: conditions — Spinal Cord Injuries; Pressure Ulcer; Motor Activity | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention, telemedicine and multidisciplinary cooperation (Experimental): The intervention group will be offered regular multidisciplinary outpatient follow-up via telemedicine.
  Interventions: Other: Service innovation with focus on multidisciplinary collaboration
- Control, multidisciplinary guidance on request. (Active Comparator): The control group will receive guidance based on existing routines (on-site consultations at the wound clinic and telephone consultations), and based on initiative taken by the local healthcare service/ patient/ next of kin.
  Interventions: Other: Service innovation with focus on multidisciplinary collaboration

INTERVENTIONS:
Other: Service innovation with focus on multidisciplinary collaboration — The follow-up is performed via telemedicine (videoconference) to the patient in his or her own home, and in cooperation with the district nurses.
  Other Names: Telemedicine in outpatient follow-up

SUMMARY:
The goal of the project is to study whether multidisciplinary follow- up performed via telemedicine to the patient in his or her own home, will improve the healthcare services offered to a particular group of patients. The hypotheses are that this could increase the treatment options, increase knowledge translation, give significant socioeconomic benefits, and allow greater accessibility to specialized healthcare services, as well as increase the involvement of patients and those working in primary healthcare.

DETAILED DESCRIPTION:
The goals of rehabilitation are to improve functional level, decrease secondary morbidity and enhance health-related quality of life. The costs associated with pressure injury are considerable. In addition to direct treatment- related costs, pressure injury also impact the hospital performance metrics. On top of the financial implications, pressure injury have a significant impact on patient morbidity and -mortality, as well as on health related quality of life. The researchers believe there is a large potential for improvement in treatment of pressure injuries. An multidisciplinary approach, including home-based rehabilitation programs, might help prevent pressure injuries and their complications, and thus reduce associated costs. The investigators conducted a pilot in 2012, in which patients with spinal cord injury and pressure injury were monitored through multidisciplinary outpatient home care, using telemedicine. The project was beneficial for the consumers/ patients, especially in terms of consumer- participation and -contribution, improved quality of life, and a better cooperation between primary and specialized healthcare services. Retrospective economic analysis indicated that telemedicine provides great savings for public healthcare services, and that using telemedicine with other patient groups with similar problems, could be beneficial. A positive outcome of the current study can be made available to most people with pressure injury. Knowledge about pressure injury will contribute in both planning and establishment of good treatment lines for the patients, as well as contribute to environmental savings, and more proper use of the health resources. This may reduce the consumption of hospital services, because a larger proportion of services are provided by the municipality. An important scientific significance of this research will thus be to improve, simplify and streamline health care and health- related services.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic or non- traumatic SCI and ongoing pressure injury.
* Consent to participate.

Exclusion Criteria:

* Patients who are unable to give their consent due to cognitive problems.
* Patients who do not have a permanent/ known address.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Health related quality of life | 1 year
  Measured by the use of SF-36, EQ-5D and SCI QoL BDS
Wound healing | 1 year
  The reduction of pressure injury size will be measured in percentage and time to healing as days from baseline to healing
Cost-utility | 1 year
  Measured in Euro, by use of QUALYs and ICER in a CE plane

SECONDARY OUTCOMES:
Experienced interaction, satisfaction and safety in the follow-up | 1 year
  Measured by use of a custom made Likert scale with 1 being completely dissatisfied and 5 being totally satisfied
Environmental evaluation | 1 year
  Measured in terms of travel distance, travel time used and travel costs by use of The Michelin Travel's Route Planner. Environmental emission due to the travel will be measured in terms of Carbon Oxide values, called CO2 equivalents

CONTACTS AND LOCATIONS:
Overall Officials: Johan K Stanghelle, Prof. MD/PhD, Study Director — University of Oslo
Locations (1):
- Sunnaas Rehabilitation Hospital, Nesoddtangen, Akershus, Norway

REFERENCES:
- [Derived] Irgens I, Kleven L, Midelfart-Hoff J, Jelnes R, Alexander M, Stanghelle JK, Rekand T. Cost-utility analysis and impact on the environment of videoconference in pressure injury. A randomized controlled trial in individuals with spinal cord injury. Spinal Cord Ser Cases. 2024 Mar 8;10(1):10. doi: 10.1038/s41394-024-00621-w. PMID 38459049
- [Derived] Irgens I, Midelfart-Hoff J, Jelnes R, Alexander M, Stanghelle JK, Thoresen M, Rekand T. Videoconferencing in Pressure Injury: Randomized Controlled Telemedicine Trial in Patients With Spinal Cord Injury. JMIR Form Res. 2022 Apr 19;6(4):e27692. doi: 10.2196/27692. PMID 35438645
- [Derived] Irgens I, Hoff JM, Sorli H, Haugland H, Stanghelle JK, Rekand T. Hospital based care at home; study protocol for a mixed epidemiological and randomized controlled trial. Trials. 2019 Jan 24;20(1):77. doi: 10.1186/s13063-019-3185-y. PMID 30678710
- See also: Protocol of the study — http://doi.org/10.1186/s13063-019-3185-y
- See also: Pressure injury occurence in people with a newly aqcuired spinal cord injury in acute care rehabilitation — http://doi.org/10.1038/s41393-020-0465-z